CLINICAL TRIAL: NCT02010801
Title: Evaluation of Tumor Ablation Effects by Irreversible Electroporation for Patients With Malignant Liver Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201010036D
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Malignant Liver Tumors
Keywords: hepatocellular carcinoma; irreversible electroporation; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IRE for tumor before tumor resection (Experimental)
  Interventions: Procedure: irreversible electroporation; Device: nanoknife AngioDynamics US Ltd

INTERVENTIONS:
Procedure: irreversible electroporation
  Other Names: nanoknife
Device: nanoknife AngioDynamics US Ltd

SUMMARY:
Liver cancer including primary hepatocellular carcinoma (HCC) and metastatic liver cancers is one the most common malignancies in the world. Over 10000 new cases per year are diagnosed in Taiwan. Despite the many treatment options, the prognosis of HCC remains dismal. More than 8000 people died of this cancer every year in Taiwan. A majority (70%to 85%) of patients present with advanced or unresectable disease. In contrast, small liver cancers can be cured with an appreciable frequency. Five-year disease-free survival exceeding 50% has been reported for surgical resection, and for the inoperable patients who do not have vascular invasion or extrahepatic spread. Radiofrequency ablation (RFA) is recommended as an alternative curative therapy. However, the main drawback of RFA is its limitation to tumor size and location. The tumors larger than 5 cm in diameter or located adjacent to vessels, could not be ablated completely.

Irreversible electroporation (IRE), developed and manufactured by AngioDynamics US Ltd, can ablate tumor by fenestrating the cancer cell membrane by electric pulse. The anti-tumor effect does not result from thermotherapy, so is also not diminished by adjacent vessels. Several pre-clinical studies have already demonstrated IRE is a safe and effective treatment for live cancers. The system has received CE mark approval in 2008 and FDA approval in 2010. However, there is no experience in using IRE fro tumor ablation in Taiwan. In this study, the investigators will perform intraoperative IRE for the patients with liver cancers who are scheduled to receive hepatectomy in our hospital, and the investigators will evaluate the ablate effect of tumors on specimens, and the effect of adjacent vessels. The investigators will appraisal the clinical feasibility and advantage of the system by this study.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC or other cancers with hepatic metastatic with pathologic proven.
* The diagnosis of HCC will be made by pathology / cytology or according to the AASLD(2010) diagnostic criteria. In brief, Nodules larger than 1 cm found on ultrasound screening of a cirrhotic liver should be investigated further with either 4-phase multidetector CT scan or dynamic contrast enhanced MRI. If the appearances are typical of HCC (i.e., hypervascular in the arterial phase with washout in the portal venous or delayed phase), the lesion should be treated as HCC. If the findings are not characteristic or the vascular profile is not typical, a second contrast enhanced study with the other imaging modality should be performed, or the lesion should be biopsied. Biopsies of small lesions should be evaluated by expert pathologists. Tissue that is not clearly HCC should be stained with all the available markers including CD34, CK7, glypican 3, HSP-70, and glutamine synthetase to improve diagnostic accuracy.
* Suitable for surgical resection, but the distance between tumors and preserved vessels is less than 5 mm. Adequate safe margin can not be obtained.
* There are at least one tumor, but less than or equal to 3 tumors,
* Each tumor must be ≤ 5 cm in diameter,
* Child-Pugh class A-B,
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* American Society of Anaesthesiologists (ASA) score ≤ 3,
* Platelet count ≥ 100 K/Μl
* Total bilirubin ≦ 2 mg/dL
* ALT and AST < 5 x upper limit of normal
* PT-INR ≦ 2.0, or PT < 6 seconds above control
* Serum creatinine ≦ 1.5 x upper limit of normal
* Prior Informed Consent Form
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Congestive heart failure >New York Heart Association (NYHA) class 2
* Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed)
* Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 3.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker
* Uncontrolled hypertension
* Any active metal implanted device (eg Pacemaker),
* Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception,
* Received treatment with an investigational agent/ procedure within 30 days prior to treatment with the NanoKnife™ IRE System,
* Known history of HIV infection
* Concurrent primary extrahepatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Complete treatment | 1 month later

SECONDARY OUTCOMES:
adverse effect | one month

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan